CLINICAL TRIAL: NCT05882396
Title: Efficacy of Rood's Approach on Oxaliplatin-induced Peripheral Neuropathy in Colorectal Cancer Patients
Brief Title: Rood's Approach and Oxaliplatin-induced Peripheral Neuropathy in Colorectal Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Ahmed Elsayeh, Lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004322
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer; Peripheral Neuropathy
Keywords: Rood's approach; Oxaliplatin-induced peripheral neuropathy; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Sixty Patients with colorectal cancer have oxaliplatin-induced peripheral neuropathy. will be indiscriminately assigned to two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rood's approach group (Active Comparator): Thirty colorectal cancer patients have oxaliplatin-induced peripheral neuropathy.
  Interventions: Other: Rood's approach; Other: Traditional physical therapy program
- Traditional physical therapy program group (Active Comparator): Thirty colorectal cancer patients have oxaliplatin-induced peripheral neuropathy.
  Interventions: Other: Traditional physical therapy program

INTERVENTIONS:
Other: Rood's approach — Patients will receive Rood's approach includes various facilitatory and inhibitory techniques.
  Arms: Rood's approach group
Other: Traditional physical therapy program — Participants will be engaged in aerobic exercises and balance training, three times per week for twelve weeks.

SUMMARY:
Oxaliplatin-induced chronic peripheral neuropathy is of major concern to oncologists and patients as it has been shown to affect patients' health-related quality of life. Although a number of interventions have been implicated, none of them can be recommended for clinical use. This therapeutic failure reflects a poor understanding of the real mechanism of oxaliplatin-induced neuropathy. However, oxidative stress is identified to be one of the main biomolecular dysfunctions in this neuropathy. Rood's approach is a neurophysiological approach that is based on reflexes of the central nervous system in which the sensory stimulation provides desired muscular response and was specially designed for patients with motor control problems. It was developed by Margeret Rood in 1940. According to Rood, sensory stimulation can activate or deactivate the receptor by facilitation or inhibition, which makes it possible to get the desired muscular response.

DETAILED DESCRIPTION:
So, the purpose of the study is to investigate the efficiency of Rood's approach on oxaliplatin-induced peripheral neuropathy in colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient can participate in the study if they had at least one cycle of oxaliplatin chemotherapy.
* Colorectal cancer patients who have oxaliplatin-induced peripheral neuropathy, the patients included in the study with mild to moderate neuropathy according to mTNS.
* Patients from both genders.
* Their ages range from 18 to 60 years old.

Exclusion Criteria:

* Patients who had a history of any other neuropathy as diabetic neuropathy.
* Patients with an unstable medical condition during chemotherapy.
* Patients who are starting new therapy or dose modification during the study period.
* Patients with morbid obesity "body mass index >40%".
* Patients with a history of non-surgically repaired nerve compression injuries such as carpal tunnel, brachial plexopathy, spinal stenosis, and spinal nerve root compression.
* Patients with a history of central nervous system primary or metastatic malignancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-12-28 (Estimated); Study Completion 2024-01-11 (Estimated)

PRIMARY OUTCOMES:
NCT-CTCAE peripheral neuropathy grading | Change from baseline at twelve weeks after the intervention
  It consists of of 5 grades; Grade (1) is asymptomatic may be accompanied by loss of tendon reflex or paraesthesia. Grade (2) is moderate symptoms which limit instrumental activities of daily life Grade (3) is severe symptoms which limit self-care activates of daily life. Grade (4) is life threatening consequences or urgent intervention indicated. Grade (5) is death.
The Ntx-12 questionnaire | Change from baseline at twelve weeks after the intervention
  It is comprised of 12 statements intended to measure the severity and impact of peripheral sensory neuropathy on patients' lives. Patients were instructed to complete the Arabic version of the Ntx-12 and choose the number corresponding to how true each statement was for them using a Likert-type scale, with 0 indicating not at all; 1, a little bit; 2, somewhat; 3, quite a bit; and 4, very much.
Brief Pain Inventory Short Form (BPI-SF) Bworst pain | Change from baseline at twelve weeks after the intervention
  The BPI-SF assesses pain at its worst, least, average, and now (current pain). Patients respond on 0-to-10 numerical rating scales. Each scale presented as a row of equidistant numbers, where 0 = no pain^ and 10 = pain as bad as you can imagine.
Total Neuropathy Score | Change from baseline at twelve weeks after the intervention
  used to measure these constructs. It includes 6 items graded from 0 to 4 according to the patients' symptoms, the total grade from 0 to 24. The higher grade the worse neuropathy. It graded as mild (1:9), moderate (10:19) and (20:24) severe.

SECONDARY OUTCOMES:
The 4-Stage Balance Test | Change from baseline at twelve weeks after the intervention
  is a recommended measure from the Centers for Disease Control and Prevention STEADI (Stopping Elderly Accidents, Deaths, and Injuries) falls campaign to recognize fall risk. An adult who cannot hold tandem stance for 10 seconds is at a higher risk for falls. [18] Patient A was able to stand in tandem stance for 2 seconds on each side. Patient B was able to stand on single leg stance for 10 seconds on each side

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa MA El Sayeh, PhD, Principal Investigator — Lecturer at Faculty of Physical Therapy, Cairo University

IPD SHARING:
Plan to Share IPD: No